CLINICAL TRIAL: NCT01667744
Title: Citalopram for Sx/Util in Acute Coronary Syndrome Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: unfunded
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Mark W. Ketterer, PhD, Senior Bioscientific Staff, Henry Ford Health System
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11146121
Record Dates: First submitted 2012-08-12; First posted 2012-08-17 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Acute Coronary Syndrome
Keywords: Angina; Acute Coronary Syndrome; Emotional Distress; Citalopram; Health Care Utilization
MeSH Terms: conditions — Acute Coronary Syndrome; Angina Pectoris; Patient Acceptance of Health Care | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo pill
  Interventions: Drug: Citalopram
- Citalopram (Experimental): Drug
  Interventions: Drug: Citalopram

INTERVENTIONS:
Drug: Citalopram — 10 mg/day

SUMMARY:
Symptoms (chest pain, shortness of breath, dizziness, etc.) and treatment usage (doctor or emergency room visits, testing, hospital days, etc.) in patients with Acute Coronary Syndromes are known to be related to emotional distress (Anxiety, Depression and Anger). In addition, behavioral treatment of emotional distress is known to decrease symptoms, and treatment usage. The present protocol tests whether the addition of a medication known to reduce emotional distress can also reduce symptoms and treatment usage.

This will done by recruiting patients with ACS during their hospital stay, randomizing them to receive citalopram or placebo, and then examining their symptoms and treatment usage at 6 months.

DETAILED DESCRIPTION:
Not applicable. Study not funded.

ELIGIBILITY:
Inclusion Criteria:

* Admission to hospital for chest pain/dyspnea, typical ECG changes plus positive tropinins

Exclusion Criteria:

* age less than 18
* cognitive impairment (per MMSE)
* geographic unavailability for followup
* unwillingness to participate
* illiteracy
* Hx cardiac transplant
* untreated hypothyroidism
* hepatic dysfunction
* prior adverse reaction to citalopram
* history of Bipolar Disorder
* untreated Sleep Apnea
* chronic steroid therapy
* active substance abuse (e.g., within past year)
* near term mortal illness
* current mental health treatment
* signitificant suicide risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01-01 (Estimated); Primary Completion 2016-02-01 (Estimated); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Frequency of ACS Symptoms | 6 months
  Frequency of episiodes of chest pain, presyncope, dyspnea, fatigue and palpitations
Treatment usage | 6 months
  ER Visits, Hospital Days, Catheterizations, PTCAs/CABGs, Valve Surgery, AICD/Pacemaker, Treadmills, Echos, Nuclear Scans, Chest X-Rays

SECONDARY OUTCOMES:
Emotional Distress | 6 months
  Depression per PHQ9, Anxiety per GAD7 & Anxiety/Depression/AIAI per KSSFC

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Ketterer, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
Study not funded.